CLINICAL TRIAL: NCT06085027
Title: Compare the Epifaith® Syringe With the Plastic Syringe for Identification of the Epidural Space in Parturients: A Prospective Randomized Control Study
Brief Title: Comparison of the Epifaith® Syringe With the Plastic Syringe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202301331A3
Record Dates: First submitted 2023-10-11; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Epidural; Anesthesia, Headache; Analgesia
MeSH Terms: conditions — Headache; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Epifaith® syringe (Experimental)
  Interventions: Procedure: Labor analgesia
- The plastic syringe (Active Comparator)
  Interventions: Procedure: Labor analgesia

INTERVENTIONS:
Procedure: Labor analgesia — Perform epidrual analgesia for parturients between 18 to 45 year-old

SUMMARY:
The goal of this clinical trial is to compare the efficiency of identifying epidural space with either the Epifaith® syringe or the plastic syringe in parturients. The main questions it aims to answer are:

* Whether it consume less time identifying epidural space with the Epifaith® syringe
* Whether the usage of the Epifaith® syringe decrease the complication rate and failure of labor analgesia Participants will receive labor analgesia either with the Epifaith® syringe or the plastic syringe conducted by experienced resident doctors.

ELIGIBILITY:
Inclusion Criteria:

* ASA II to III
* Require labor analgesia
* Has submitted inform consent

Exclusion Criteria:

* ASA IV or above
* Coagulopathy
* Spinal deformity
* Neurological, psychological, cardiopulmonary disorder
* Active liver or kidney injury

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Time consumed to identify the epidural space | During the procedure
  Starting on the moment which the syringe be attached to the needle